CLINICAL TRIAL: NCT01914757
Title: A Multicentre, Randomized, Double-blind, Parallel Group, Placebocontrolled, Phase 3 Study to Evaluate the Efficacy and Safety of Benralizumab in Asthmatic Adults and Adolescents Inadequately Controlled on Inhaled Corticosteroid Plus Long-acting β2 Agonist (CALIMA)
Brief Title: Efficacy and Safety Study of Benralizumab in Adults and Adolescents Inadequately Controlled on Inhaled Corticosteroid Plus Long-acting β2 Agonist
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3250C00018
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Results first posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: Asthma, Bronchial Diseases, Respiratory Tract Diseases, Lung Diseases, Obstructive Lung Diseases
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Benralizumab 30 mg q.4 weeks (Experimental): Benralizumab administered subcutaneously every 4 weeks
  Interventions: Biological: Benralizumab
- Benralizumab 30 mg q.8 weeks (Experimental): Benralizumab administered subcutaneously every 8 weeks
  Interventions: Biological: Benralizumab
- Placebo (Placebo Comparator): Placebo administered subcutaneously
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Benralizumab — Benralizumab subcutaneously on study week 0 until study week 52 inclusive.
  Arms: Benralizumab 30 mg q.4 weeks; Benralizumab 30 mg q.8 weeks
Biological: Placebo — Placebo subcutaneously on study week 0 until study week 52 inclusive.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Benralizumab reduces the exacerbation rate in patients with a history of asthma exacerbations and uncontrolled asthma receiving ICS-LABA with or without oral corticosteroids and additional asthma controllers.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female and male aged 12 to 75 years, inclusively, at the time of Visit 1
3. History of physician-diagnosed asthma requiring treatment with medium-to-high dose ICS (>250µg fluticasone dry powder formulation equivalents total daily dose) and a LABA, for at least 12 months prior to Visit 1.
4. Documented treatment with ICS and LABA for at least 3 months prior to Visit 1 with or without oral corticosteroids and additional asthma controllers. The ICS and LABA can be parts of a combination product or given by separate inhalers. The ICS dose must be greater than or equal to 500 μg/day fluticasone propionate dry powder formulation or equivalent daily. For ICS/LABA combination preparations, the mid-strength approved maintenance dose in the local country will meet this ICS criterion.

Exclusion criteria:

1. Clinically important pulmonary disease other than asthma (e.g. active lung infection, COPD, bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha 1 anti-trypsin deficiency, and primary ciliary dyskinesia) or ever been diagnosed with pulmonary or systemic disease, other than asthma, that are associated with elevated peripheral eosinophil counts (e.g. allergic bronchopulmonary aspergillosis/mycosis, Churg- Strauss syndrome, hypereosinophilic syndrome)
2. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could:

   * Affect the safety of the patient throughout the study
   * Influence the findings of the studies or their interpretations
   * Impede the patient's ability to complete the entire duration of study
3. Acute upper or lower respiratory infections requiring antibiotics or antiviral medication within 30 days prior to the date informed consent is obtained or during the screening/run-in period
4. Any clinically significant abnormal findings in physical examination, vital signs, haematology, clinical chemistry, or urinalysis during screening/run-in period, which in the opinion of the Investigator, may put the patient at risk because of his/her participation in the study, or may influence the results of the study, or the patient's ability to complete entire duration of the study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2508 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fitzgerald, MD, PhD, Professor of Medicine, Principal Investigator — The Lung Centre, Gordon and Leslie Diamond Health Care Centre, Vancouver Canada
Locations (215):
- United States (81):
  - Research Site, Andalusia, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Flagstaff, Arizona
  - Research Site, Glendale, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Alhambra, California
  - Research Site, Anaheim, California
  - Research Site, Beverly Hills, California
  - Research Site, Garden Grove, California
  - Research Site, Lakewood, California
  - Research Site, North Hollywood, California
  - Research Site, Northridge, California
  - Research Site, Palmdale, California
  - Research Site, Rancho Mirage, California
  - Research Site, Redondo Beach, California
  - Research Site, Rolling Hills Estate, California
  - Research Site, Sacramento, California
  - Research Site, Stockton, California
  - Research Site, Thousand Oaks, California
  - Research Site, Upland, California
  - Research Site, Ventura, California
  - Research Site, Walnut Creek, California
  - Research Site, Westminster, California
  - Research Site, Woodland, California
  - Research Site, Centennial, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Celebration, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Homestead, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lehigh Acres, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Virginia Gardens, Florida
  - Research Site, Gainesville, Georgia
  - Research Site, Smyrna, Georgia
  - Research Site, Eagle, Idaho
  - Research Site, Shiloh, Illinois
  - Research Site, Lenexa, Kansas
  - Research Site, Fort Mitchell, Kentucky
  - Research Site, Covington, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Farmington Hills, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Traverse City, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Las Vagas, Nevada
  - Research Site, Union, New Jersey
  - Research Site, The Bronx, New York
  - Research Site, Durham, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Corvallis, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Jefferson Hills, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Old Point Station, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Knoxville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Boerne, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Midvale, Utah
  - Research Site, Murray, Utah
  - Research Site, Fairfax, Virginia
  - Research Site, Falls Church, Virginia
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Argentina (15):
  - Research Site, Buenos Aires
  - Research Site, Caba
  - Research Site, Ciudad Autónoma de Bs. As.
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Concepción del Uruguay
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Florida
  - Research Site, Godoy Cruz
  - Research Site, La Plata
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Ranelagh
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
- Canada (11):
  - Research Site, Calgary, Alberta
  - Research Site, Sherwood Park, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Moncton, New Brunswick
  - Research Site, Burlington, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
- Chile (6):
  - Research Site, Concepción
  - Research Site, Quillota
  - Research Site, Santiago
  - Research Site, Talcahuano
  - Research Site, Valparaíso
  - Research Site, Viña del Mar
- Germany (18):
  - Research Site, Aschaffenburg
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Geesthacht
  - Research Site, Gelsenkirchen
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Herford
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, München
  - Research Site, Neu-Isenburg
  - Research Site, Rostock
  - Research Site, Rüdersdorf
  - Research Site, Witten
- Japan (31):
  - Research Site, Asahi-shi
  - Research Site, Chiyoda-ku
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Himeji-shi
  - Research Site, Hiroshima
  - Research Site, Itabashi-ku
  - Research Site, Kagoshima
  - Research Site, Kishiwada-shi
  - Research Site, Kobe
  - Research Site, Kokubunji-shi
  - Research Site, Matsue
  - Research Site, Minatoku
  - Research Site, Mizunami-shi
  - Research Site, Niigata
  - Research Site, Obihiro-shi
  - Research Site, Ota-shi
  - Research Site, Ōita
  - Research Site, Sagamihara-shi
  - Research Site, Sakaide-shi
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Setagaya-ku
  - Research Site, Shibuya-ku
  - Research Site, Shinagawa-ku
  - Research Site, Sumida-ku
  - Research Site, Takamatsu
  - Research Site, Toshima-ku
  - Research Site, Tsukubo-gun
  - Research Site, Yokohama
- Philippines (3):
  - Research Site, Iloilo City
  - Research Site, Lipa City
  - Research Site, Quezon City
- Poland (29):
  - Research Site, Aleksandrów Łódzki
  - Research Site, Bialystok
  - Research Site, Bielsko-Biala
  - Research Site, Bydgoszcz
  - Research Site, Bystra
  - Research Site, Gdansk
  - Research Site, Gorzów Wlkp
  - Research Site, Karczew
  - Research Site, Katowice
  - Research Site, Koszalin
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lubin
  - Research Site, Lublin
  - Research Site, Ostrów Wielkopolski
  - Research Site, Poznan
  - Research Site, Ruda Śląska
  - Research Site, Rzeszów
  - Research Site, Skierniewice
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Torun
  - Research Site, Trzebnica
  - Research Site, Warsaw
  - Research Site, Wieluń
  - Research Site, Wroclaw
  - Research Site, Zabrze
  - Research Site, Żnin
  - Research Site, Łęczna
- Romania (7):
  - Research Site, Bragadiru
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Constanța
  - Research Site, Deva
  - Research Site, Iași
  - Research Site, Timișoara
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Luleå
  - Research Site, Lund
- Ukraine (11):
  - Research Site, Chernivtsi
  - Research Site, Dnipropetrovsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Mykolayiv
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
  - Research Site, Zaporizhzhya

REFERENCES:
- [Derived] Menzies-Gow A, Hoyte FL, Price DB, Cohen D, Barker P, Kreindler J, Jison M, Brooks CL, Papeleu P, Katial R. Clinical Remission in Severe Asthma: A Pooled Post Hoc Analysis of the Patient Journey with Benralizumab. Adv Ther. 2022 May;39(5):2065-2084. doi: 10.1007/s12325-022-02098-1. Epub 2022 Mar 14. PMID 35287231
- [Derived] Lugogo NL, Kreindler JL, Martin UJ, Cook B, Hirsch I, Trudo FJ. Blood eosinophil count group shifts and kinetics in severe eosinophilic asthma. Ann Allergy Asthma Immunol. 2020 Aug;125(2):171-176. doi: 10.1016/j.anai.2020.04.011. Epub 2020 Apr 22. PMID 32334141
- [Derived] Jackson DJ, Humbert M, Hirsch I, Newbold P, Garcia Gil E. Ability of Serum IgE Concentration to Predict Exacerbation Risk and Benralizumab Efficacy for Patients with Severe Eosinophilic Asthma. Adv Ther. 2020 Feb;37(2):718-729. doi: 10.1007/s12325-019-01191-2. Epub 2019 Dec 14. PMID 31836949
- [Derived] Chipps BE, Hirsch I, Trudo F, Alacqua M, Zangrilli JG. Benralizumab efficacy for patients with fixed airflow obstruction and severe, uncontrolled eosinophilic asthma. Ann Allergy Asthma Immunol. 2020 Jan;124(1):79-86. doi: 10.1016/j.anai.2019.10.006. Epub 2019 Oct 15. PMID 31626906
- [Derived] Chupp G, Lugogo NL, Kline JN, Ferguson GT, Hirsch I, Goldman M, Zangrilli JG, Trudo F. Rapid onset of effect of benralizumab on morning peak expiratory flow in severe, uncontrolled asthma. Ann Allergy Asthma Immunol. 2019 May;122(5):478-485. doi: 10.1016/j.anai.2019.02.016. Epub 2019 Feb 23. PMID 30802500
- [Derived] Bleecker ER, Wechsler ME, FitzGerald JM, Menzies-Gow A, Wu Y, Hirsch I, Goldman M, Newbold P, Zangrilli JG. Baseline patient factors impact on the clinical efficacy of benralizumab for severe asthma. Eur Respir J. 2018 Oct 18;52(4):1800936. doi: 10.1183/13993003.00936-2018. Print 2018 Oct. PMID 30139780
- [Derived] DuBuske L, Newbold P, Wu Y, Trudo F. Seasonal variability of exacerbations of severe, uncontrolled eosinophilic asthma and clinical benefits of benralizumab. Allergy Asthma Proc. 2018 Sep 4;39(5):345-349. doi: 10.2500/aap.2018.39.4162. Epub 2018 Aug 4. PMID 30077185
- [Derived] Chipps BE, Newbold P, Hirsch I, Trudo F, Goldman M. Benralizumab efficacy by atopy status and serum immunoglobulin E for patients with severe, uncontrolled asthma. Ann Allergy Asthma Immunol. 2018 May;120(5):504-511.e4. doi: 10.1016/j.anai.2018.01.030. Epub 2018 Feb 1. PMID 29409951
- [Derived] Ohta K, Adachi M, Tohda Y, Kamei T, Kato M, Mark Fitzgerald J, Takanuma M, Kakuno T, Imai N, Wu Y, Aurivillius M, Goldman M. Efficacy and safety of benralizumab in Japanese patients with severe, uncontrolled eosinophilic asthma. Allergol Int. 2018 Apr;67(2):266-272. doi: 10.1016/j.alit.2017.10.004. Epub 2017 Nov 8. PMID 29128192
- [Derived] FitzGerald JM, Bleecker ER, Nair P, Korn S, Ohta K, Lommatzsch M, Ferguson GT, Busse WW, Barker P, Sproule S, Gilmartin G, Werkstrom V, Aurivillius M, Goldman M; CALIMA study investigators. Benralizumab, an anti-interleukin-5 receptor alpha monoclonal antibody, as add-on treatment for patients with severe, uncontrolled, eosinophilic asthma (CALIMA): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2016 Oct 29;388(10056):2128-2141. doi: 10.1016/S0140-6736(16)31322-8. Epub 2016 Sep 5. PMID 27609406
- See also: D3250C00018CSP3redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1823&filename=d3250c00018_Revised_CSP_CALIMA..pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2505 participants signed informed consent, 2181 entered screening/run-in period, 1306 participants were randomised to receive treatment with benralizumab 30 mg Q4W, Q8W, or placebo. Of the 1306 patients randomised, all (100.0%) received treatment with study drug.
Period: Overall Study
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Started | 425 | 441 | 440
Completed | 389 | 390 | 402
Not Completed | 36 | 51 | 38
Not completed — Severe non-compliance to protocol | 3 | 1 | 2
Not completed — Lost to Follow-up | 5 | 8 | 6
Not completed — Withdrawal by Subject | 15 | 27 | 19
Not completed — Death | 2 | 2 | 1
Not completed — Adverse Event | 4 | 3 | 4
Not completed — Study specific withdrawal criteria | 0 | 1 | 0
Not completed — Eligibility criteria not fulfilled | 2 | 0 | 2
Not completed — Other reasons | 5 | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo | Total
Number analyzed (Participants) | 425 | 441 | 440 | 1306
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.0 (13.6) | 49 (14.3) | 48.8 (15.1) | 49.2 (14.3)
Gender [Count of Participants; unit: Participants]
  Female | 270 | 273 | 264 | 807
  Male | 155 | 168 | 176 | 499

OUTCOME MEASURES:

1. Primary Outcome: Annual Asthma Exacerbation Rate in Adult and Adolescent Patients With Uncontrolled Asthma for Patients With Baseline Eosinophils >=300/uL
Description: The annual exacerbation rate is based on unadjudicated annual exacerbation rate reported by the investigator in the eCRF.
Time Frame: Immediately following the first administration of study drug through Study Week 56.
Population: Full analysis set, Baseline eosinophils >=300/uL, High-dose ICS.
Measure: Least Squares Mean (95% Confidence Interval); unit: Events/year
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 241 | 239 | 248
Events/year | 0.6 [0.48 to 0.74] | 0.66 [0.54 to 0.82] | 0.93 [0.77 to 1.12]
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.002, Negative Binomial; Model includes covariates treatment group, region, number of exacerbations in the previous year, and use of maintenance oral corticosteroids; Rate Ratio = 0.64, 95% CI 2-sided [0.49 to 0.85]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.019, Negative Binomial; [statistical method as in outcome 1, analysis 1]; Rate Ratio = 0.72, 95% CI 2-sided [0.54 to 0.95]

2. Secondary Outcome: Annual Asthma Exacerbation Rate in Adult and Adolescent Patients With Uncontrolled Asthma for Patients With Baseline Eosinophils <300/uL
Description: as for outcome 1
Time Frame: Immediately following the first administration of study drug through Study Week 56.
Population: Full analysis set, Baseline eosinophils <300/uL, High-dose ICS.
Measure: Least Squares Mean (95% Confidence Interval); unit: Events/year
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 116 | 125 | 122
Events/year | 0.78 [0.59 to 1.02] | 0.73 [0.55 to 0.95] | 1.21 [0.96 to 1.52]
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.015, Negative Binomial; [statistical method as in outcome 1, analysis 1]; Rate Ratio = 0.64, 95% CI 2-sided [0.45 to 0.92]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.005, Negative Binomial; [statistical method as in outcome 1, analysis 1]; Rate Ratio = 0.6, 95% CI 2-sided [0.42 to 0.86]

3. Secondary Outcome: Mean Change From Baseline to Week 56 in Pre-bronchodilator FEV1 (L) Value for Patients With Baseline Eosinophils >=300/uL
Time Frame: Immediately following the first administration of study drug through Study Week 56.
Population: Full analysis set, Baseline eosinophils >=300/uL, High-dose ICS
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 216 | 211 | 221
Liter | 0.34 (0.469) | 0.332 (0.518) | 0.206 (0.471)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; Model includes treatment, baseline pre-BD FEV1, region, use of OCS, visit, and treatment by visit; Mean Difference (Final Values) = 0.125, 95% CI 2-sided [0.037 to 0.213]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis; Model includes treatment, baseline pre-BD FEV1, region, use of OCS, visit, and treatment by visit; Mean Difference (Final Values) = 0.116, 95% CI 2-sided [0.028 to 0.204]

4. Secondary Outcome: Mean Change From Baseline to Week 56 in Pre-bronchodilator FEV1 (L) Value for Patients With Baseline Eosinophils <300/uL
Time Frame: Immediately following the first administration of study drug through Study Week 56.
Population: Full analysis set, Baseline eosinophils <300/uL, High-dose ICS
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 101 | 98 | 99
Liter | 0.221 (0.441) | 0.164 (0.358) | 0.135 (0.437)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.268, Mixed Models Analysis; Model includes treatment, baseline pre-BD FEV1, region, use of OCS, visit, and treatment by visit; Mean Difference (Final Values) = 0.064, 95% CI 2-sided [-0.049 to 0.176]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.786, Mixed Models Analysis; Model includes treatment, baseline pre-BD FEV1, region, use of OCS, visit, and treatment by visit; Mean Difference (Final Values) = -0.015, 95% CI 2-sided [-0.127 to 0.096]

5. Secondary Outcome: Mean Change From Baseline to Week 56 Asthma Symptoms Score for Patients With Baseline Eosinophils >=300/uL
Description: Asthma symptoms during night time and daytime are recorded by the patient each morning and evening in the asthma daily diary. Symptom score values are from 0 (No asthma symptom) to 3 (unable to sleep because of asthma). Baseline is defined as the average of data collected from the evening of study day -10 to the morning of study day 1. Each timepoint is calculated as bi-weekly means based on daily diary data. If more than 50% of scores are missing in a 14 day period then this is considered as missing. Symptom score lower is better.
Time Frame: Immediately following the first administration of study drug through Study Week 56.
Population: Full analysis set, Baseline eosinophils >=300/uL, High-dose ICS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 184 | 185 | 187
Scores on a scale | -1.33 (1.23) | -1.4 (1.17) | -1.2 (1.19)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.224, Mixed Models Analysis; Model includes treatment, baseline Asthma symptom score, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.32 to 0.07]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis; Model includes treatment, baseline Asthma symptom score, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.43 to -0.04]

6. Secondary Outcome: Mean Change From Baseline to Week 56 Asthma Symptoms Score for Patients With Baseline Eosinophils <300/uL
Description: as for outcome 5
Time Frame: Immediately following the first administration of study drug through Study Week 56.
Population: Full analysis set, Baseline eosinophils <300/uL, High-dose ICS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 88 | 85 | 89
Scores on a scale | -1.05 (1.14) | -0.95 (1.13) | -0.88 (1.12)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.287, Mixed Models Analysis; Model includes treatment, baseline Asthma symptom score, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.44 to 0.13]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.966, Mixed Models Analysis; Model includes treatment, baseline Asthma symptom score, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.28 to 0.29]

7. Secondary Outcome: Change in Asthma Rescue Medication Use
Description: Change from Baseline to Week 56 in number of Rescue medication use (puffs/day)
Time Frame: Immediately following the first administration of study drug through Study Week 56.
Population: Full analysis set, Baseline eosinophils >=300/uL, High-dose ICS
Measure: Mean (Standard Deviation); unit: Puffs per day
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 184 | 185 | 187
Puffs per day | -2.0 (3.64) | -2.92 (3.60) | -2.65 (9.57)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.603, Mixed Models Analysis; Model includes treatment, baseline Asthma rescue medication use, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.58 to 0.99]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.209, Mixed Models Analysis; Model includes treatment, baseline Asthma medication use, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.29 to 0.28]

8. Secondary Outcome: Home Lung Function Assessments Based on PEF
Description: Change from Baseline to Week 56 in Home lung function (morning and evening Peak expiratory flow [PEF])
Time Frame: Immediately following the first administration of study drug through Study Week 56.
Population: Full analysis set, Baseline eosinophils >=300/uL, High-dose ICS
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 241 | 239 | 248
L/min
  Change at Week 56, Morning (n=194, 193, 197) | 41.745 (78.534) | 43.375 (91.865) | 23.961 (71.509)
  Change at Week 56, Evening (n=194, 192, 197) | 35.142 (75.489) | 39.270 (89.772) | 15.448 (78.341)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Morning PEF Change from Baseline to Week 56; Test type: Superiority or Other; p = 0.029, Mixed Models Analysis; Model includes treatment, baseline morning PEF, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = 15.86, 95% CI 2-sided [1.59 to 30.12]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Morning PEF Change from Baseline to Week 56; Test type: Superiority or Other; p = 0.037, Mixed Models Analysis; Model includes treatment, baseline morning PEF, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = 15.27, 95% CI 2-sided [0.9 to 29.64]
Statistical Analysis 3: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Evening PEF Change from Baseline to Week 56; Test type: Superiority or Other; p = 0.018, Mixed Models Analysis; Model includes treatment, baseline evening PEF, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = 17.54, 95% CI 2-sided [3.07 to 32]
Statistical Analysis 4: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Evening PEF Change from Baseline to Week 56; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Model includes treatment, baseline evening PEF, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = 21.22, 95% CI 2-sided [6.65 to 35.79]

9. Secondary Outcome: Proportion of Nights With Awakening Due to Asthma
Description: Change from Baseline to Week 56 on Proportion of Nights with awakening due to asthma
Time Frame: Immediately following the first administration of study drug through Study Week 56.
Population: Full analysis set, Baseline eosinophils >=300/uL, High-dose ICS
Measure: Mean (Standard Deviation); unit: Proportion of nights
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 196 | 198 | 203
Proportion of nights | -0.373 (0.388) | -0.431 (0.4) | -0.372 (0.405)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.4, Mixed Models Analysis; Model includes treatment, baseline prop of nights with nocturnal wakening, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.06 to 0.03]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.146, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.08 to 0.01]

10. Secondary Outcome: Mean Change From Baseline to Week 56 in ACQ-6 for Patients With Baseline Eosinophils >=300/uL
Description: ACQ-6 contains one bronchodilator question and 5 symptom questions. Questions are rated from 0 (totally controlled) to 6 (severely uncontrolled). Mean ACQ-6 score is the average of the responses. Mean scores of <=0.75 indicates well-controlled asthma, scores between 0.75 to <=1.5 indicate partly controlled asthma, and >1.5 indicates not well controlled asthma.
Time Frame: Immediately following the first administration of study drug through Study Week 56.
Population: Full analysis set, Baseline eosinophils >=300/uL, High-dose ICS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 192 | 185 | 197
Scores on a scale | -1.34 (1.13) | -1.49 (1.13) | -1.21 (1.12)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.043, Mixed Models Analysis; Model includes treatment, baseline ACQ-6 score, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.38 to -0.01]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis; Model includes treatment, baseline ACQ-6 score, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.44 to -0.07]

11. Secondary Outcome: Mean Change From Baseline to Week 56 in ACQ-6 for Patients With Baseline Eosinophils <300/uL
Description: as for outcome 10
Time Frame: Immediately following the first administration of study drug through Study Week 56.
Population: Full analysis set, Baseline eosinophils <300/uL, High-dose ICS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 88 | 83 | 92
Scores on a scale | -1.22 (1.16) | -1.06 (1.02) | -0.83 (1.07)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.078, Mixed Models Analysis; Model includes treatment, baseline ACQ-6 score, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.51 to 0.03]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.449, Mixed Models Analysis; Model includes treatment, baseline ACQ-6 score, region, use of OCS, visit, and visit by treatment; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.37 to 0.16]

12. Secondary Outcome: Number of Patients With >=1 Asthma Exacerbation
Time Frame: Immediately following the first administration of study drug through Study Week 56
Population: Full analysis set, Baseline eosinophils >=300/uL, High-dose ICS
Measure: Number; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 241 | 239 | 248
Participants | 84 | 95 | 126
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Proportion of patients with >=1 asthma exacerbation; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for region, number of exacerbations in the previous year, use of OCS; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.31 to 0.69]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Proportion of patients with >=1 asthma exacerbation; Test type: Superiority or Other; p = 0.023, Cochran-Mantel-Haenszel; Controlling for region, number of exacerbations in the previous year, use of OCS; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.45 to 0.95]

13. Secondary Outcome: Time to First Asthma Exacerbation
Time Frame: Immediately following the first administration of study drug through Study Week 56
Population: Full analysis set, Baseline eosinophils >=300/uL, High-dose ICS
Measure: Number; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 241 | 239 | 248
Participants | 84 | 95 | 126
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Time to first Exacerbation; Test type: Superiority or Other; p < 0.001, Regression, Cox; Model includes treatment, region, number of exacerbations in the previous year, use of OCS; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.46 to 0.80]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Time to first asthma exacerbation; Test type: Superiority or Other; p = 0.018, Regression, Cox; Model includes treatment, region, number of exacerbations in the previous year, use of OCS; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.55 to 0.95]

14. Secondary Outcome: Annual Rate of Asthma Exacerbation Resulting Emergency Room Visits and Hospitalizations
Description: Annual rate of asthma exacerbations that are associated with an emergency room visit or a hospitalization (adjudicated)
Time Frame: Immediately following the first administration of study drug through Study Week 56.
Population: Full analysis set, Baseline eosinophils >=300/uL, High-dose ICS
Measure: Least Squares Mean (95% Confidence Interval); unit: Events/year
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 241 | 239 | 248
Events/year | 0.04 [0.02 to 0.06] | 0.05 [0.03 to 0.08] | 0.04 [0.02 to 0.07]
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.837, negative binomial; Model includes treatment, region, any prior exacerbation resulting ER/Hospitalization, use of OCS; Rate Ratio = 0.93, 95% CI 2-sided [0.48 to 1.82]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.538, negative binomial; Model includes treatment, region, any prior exacerbation resulting ER/Hospitalization, use of OCS; Rate Ratio = 1.23, 95% CI 2-sided [0.64 to 2.35]

15. Secondary Outcome: Pharmacokinetics of Benralizumab
Description: Mean PK Concentration at each visit
Time Frame: Baseline, Week 4, Week 8, Week 16, Week 24, Week 32, Week 40, Week 48, Week 56, Week 60
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 435 | 424 | 0
ng/mL
  Baseline (n=435, 419) | NA (NA) — Value is less than lower limit of quantification | NA (NA) — Value is less than lower limit of quantification |
  Week 4 (n=430, 416) | 650.04 (154.61) | 703.16 (89.48) |
  Week 8 (n=414, 395) | 894.86 (148.91) | 939.45 (98.99) |
  Week 16 (n=390, 378) | 936.43 (247.46) | 252.54 (274.74) |
  Week 24 (n=388, 361) | 827.09 (370.64) | 188.99 (308.38) |
  Week 32 (n=345, 323) | 823.21 (362.43) | 166.53 (289.34) |
  Week 40 (n=370, 338) | 859.69 (364.28) | 172.28 (298.6) |
  Week 48 (n=355, 337) | 888.09 (333.98) | 186.5 (290.28) |
  Week 56 (n=358, 344) | 763.98 (309.18) | 173.41 (235.86) |
  Week 60 (n=49, 45) | 53.63 (1782.96) | 18.63 (756.47) |

16. Secondary Outcome: Immunogenicity of Benralizumab
Description: Anti-drug antibodies (ADA) responses at baseline and post baseline. Persistently positive is defined as positive at >=2 post-baseline assessments (with >=16 weeks between first and last positive) or positive at last post-baseline assessment. Transiently positive is defined as having at least one post-baseline ADA positive assessment and not fulfilling the conditions of persistently positive.
Time Frame: Pre-treatment until end of follow-up
Population: Safety analysis set
Measure: Number; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 438 | 427 | 440
Participants
  Positive at any visit (n=438, 427, 440) | 63 | 64 | 13
  Base- and Post-baseline Postive (n=431, 414, 430) | 5 | 5 | 5
  Only post-baseline positive (n=431, 420, 436) | 55 | 57 | 8
  Persistently positive (n=431, 420, 436) | 44 | 42 | 7
  Transient positive (n=431, 420, 436) | 16 | 20 | 6
  Only baseline positive (n=438, 421, 434) | 3 | 2 | 0

17. Secondary Outcome: Extent of Exposure
Description: Extent of exposure is defined as the duration of treatment in days
Time Frame: Immediately following the first administration of study drug through Study Week 56
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 438 | 428 | 440
Days | 344.14 (73.129) | 331.64 (88.839) | 336.69 (82.148)

18. Secondary Outcome: Mean Change From Baseline to Week 56 in AQLQ(S)+12
Description: AQLQ(S)+12 overall score is defined as the average of all 32 questions in the AQLQ(S)+12 questionnaire. AQLQ(S)+12 is a 7-point scale questionnaire, ranging from 7 (no impairment) to 1 (severe impairment). Total or domain score change of >=0.5 are considered clinically meaningful.
Time Frame: Immediately following the first administration of study drug through Study Week 56
Population: Full analysis set, Baseline eosinophils >=300/uL, High-dose ICS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 186 | 180 | 191
Scores on a scale | 1.44 (1.15) | 1.61 (1.24) | 1.32 (1.19)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.119, Mixed Models Analysis; Model includes treatment, baseline AQLQ score, region, use of OCS, visit, visit by treatment; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.04 to 0.37]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis; Model includes treatment, baseline AQLQ score, region, use of OCS, visit, visit by treatment; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [0.04 to 0.45]

19. Secondary Outcome: Change From Baseline to Week 56 in EQ-5D-5L VAS
Description: EQ-5D-5L VAS is to rate current health status on a scale of 0-100, with 0 being the worst imaginable health state.
Time Frame: Immediately following the first administration of study drug through Study Week 56
Population: Full analysis set, Baseline eosinophils >=300/uL, High-dose ICS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 183 | 179 | 191
Scores on a scale | 13.8 (21.52) | 15.5 (20.36) | 12.1 (20.13)

20. Secondary Outcome: Mean Work Productivity Loss Due to Asthma
Description: WPAI+CIQ (Work Productivity and Activity Impairment plus Classroom Impairment Questionnaire) contains 10 questions. Work productivity loss is derived by sum of percentage of missed work due to asthma and product of percentage of actual working hours times degree of asthma affecting work productivity while working. Percentage of missed work due to asthma is calculated by number of hours missed work due to asthma divided by total number of hours missed work plus number of hours actually worked. This is only applicable to patients who were employed.
Time Frame: Immediately following the first administration of study drug through Study Week 56
Population: Full analysis set, Baseline eosinophils >=300/uL, High-dose ICS, who were employed
Measure: Mean (Standard Deviation); unit: Percent of productivity loss
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 92 | 74 | 85
Percent of productivity loss | 26.56 (25.589) | 24.44 (24.689) | 27.29 (25.802)

21. Secondary Outcome: Mean Productivity Loss Due to Asthma in Classroom
Description: WPAI+CIQ (Work Productivity and Activity Impairment plus Classroom Impairment Questionnaire) contains 10 questions. Classroom productivity loss is derived by sum of percentage of missed classes due to asthma and product of percentage of actual hours attending classes times degree of asthma affecting classroom productivity. Percentage of missed classes due to asthma is calculated by number of hours missed classes due to asthma divided by total number of hours missed classes plus number of hours actually attending classes. This is only applicable for patients who took classes.
Time Frame: Immediately following the first administration of study drug through Study Week 56
Population: Full analysis set, Baseline eosinophils >=300/uL, High-dose ICS, who took classes
Measure: Mean (Standard Deviation); unit: percent of productivity loss
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 14 | 5 | 5
percent of productivity loss | 19.92 (23.765) | 14 (16.733) | 33.5 (25.593)

22. Secondary Outcome: Number of Participants That Utilized Health Care Resources
Time Frame: Immediately following the first administration of study drug through Study Week 56
Population: Full analysis set, Baseline eosinophils >=300/uL, High-dose ICS
Measure: Number; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 241 | 239 | 248
Participants
  Hospitalizations | 11 | 14 | 12
  Emergency department visits | 11 | 12 | 18
  Unscheduled outpatient visits | 72 | 75 | 83
  Home visits | 3 | 1 | 2
  Telephone calls | 50 | 63 | 58
  Ambulance transports | 2 | 3 | 5

23. Secondary Outcome: Patient and Clinician Assessment of Response to Treatment
Description: CGIC (clinician global impression of change), and PGIC (patient global impression of change) are overall evaluation of response to treatment, conducted separately by investigator and patient using a 7-point rating scale, ranging from 1 (Very much Improved), to 7 (Very much Worse). This endpoint was added after the second protocol amendment, thus not all patients had data to be analyzed.
Time Frame: Immediately following the first administration of study drug through Study Week 56
Population: Full analysis set, Baseline eosinophils >=300/uL, High-dose ICS
Measure: Number; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 241 | 239 | 248
Participants
  CGIC, Improved | 109 | 96 | 97
  CGIC, Much Improved | 82 | 71 | 65
  CGIC, Very Much Improved | 26 | 23 | 14
  CGIC, Total | 217 | 190 | 176
  PGIC, Improved | 109 | 95 | 99
  PGIC, Much Improved | 83 | 80 | 66
  PGIC, Very Much Improved | 34 | 30 | 17
  PGIC, Total | 226 | 205 | 182

ADVERSE EVENTS:
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Serious Adverse Events (participants affected / at risk) | 46/438 | 41/428 | 61/440
Other Adverse Events (participants affected / at risk) | 244/438 | 232/428 | 264/440
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab 30 mg q.4 Weeks (N=438) | Benralizumab 30 mg q.8 Weeks (N=428) | Placebo (N=440)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus hepatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 4 (6)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0) | 3 (3)
Pseudomonas bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 21 (25) | 19 (27) | 23 (38)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Parakeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab 30 mg q.4 Weeks (N=438) | Benralizumab 30 mg q.8 Weeks (N=428) | Placebo (N=440)
Pyrexia (General disorders) | 16 (20) | 13 (13) | 6 (6)
Acute sinusitis (Infections and infestations) | 6 (6) | 5 (6) | 14 (19)
Bronchitis (Infections and infestations) | 40 (51) | 45 (54) | 54 (72)
Influenza (Infections and infestations) | 24 (27) | 12 (17) | 25 (27)
Nasopharyngitis (Infections and infestations) | 90 (132) | 82 (131) | 92 (147)
Pharyngitis (Infections and infestations) | 17 (21) | 10 (10) | 8 (9)
Rhinitis (Infections and infestations) | 12 (13) | 18 (24) | 17 (22)
Sinusitis (Infections and infestations) | 23 (31) | 21 (30) | 39 (56)
Upper respiratory tract infection (Infections and infestations) | 29 (35) | 37 (53) | 42 (53)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 14 (16) | 10 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (18) | 11 (11) | 16 (20)
Headache (Nervous system disorders) | 33 (63) | 34 (65) | 32 (57)
Asthma (Respiratory, thoracic and mediastinal disorders) | 50 (76) | 32 (50) | 52 (96)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 14 (18) | 8 (12)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 21 (25) | 16 (19) | 24 (28)
Hypertension (Vascular disorders) | 12 (12) | 18 (23) | 22 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
≥ 60 days prior to submission of material for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Inst. and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication or presentation.